CLINICAL TRIAL: NCT04338451
Title: Music Listening to Decrease Pain and Discomfort During Extracorporeal Shock Wave Lithotripsy (SWL): a Prospective Randomized Trial.
Brief Title: Music During ESWL for Half Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Andrea Bosio, Principal investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOUCSSTURAB001
Record Dates: First submitted 2015-12-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; Kidney Calculi; Lithotripsy; Pain Management; Music
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music during the first part of ESWL (Active Comparator): Patients listen to music during the first part of ESWL treatment (first 1800 SW).
  Interventions: Other: Music during the first part of ESWL
- Music during the second part of ESWL (Active Comparator): Patients listen to music during the second part of ESWL treatment.
  Interventions: Other: Music during the second part of ESWL

INTERVENTIONS:
Other: Music during the first part of ESWL — Music listening during first part of ESWL
  Arms: Music during the first part of ESWL
Other: Music during the second part of ESWL — Music listening during second part of ESWL
  Arms: Music during the second part of ESWL

SUMMARY:
The aim of this study is to evaluate if music listening relieves pain and discomfort during Extracorporeal Shock-Waves Lithotripsy (ESWL).

DETAILED DESCRIPTION:
Patients undergoing ESWL and interested in music listening are randomly divided in two groups: patients in group A listen to music during the first part of the treatment (first 1800 SW), patients in group B during the second part.

At the end of the treatment patients are asked to fill in a questionnaire. They are asked if they were pleased to have had the opportunity to listen to music during ESWL, if they would like to listen to music again in case of further treatments, if they consider music helpful in relieving pain and discomfort during ESWL. Patients are also asked to mark their level of pain during each part of the treatment on a visual analogue scale (VAS) for pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ESWL from February 2011 to October 2012 and interested in music listening

Exclusion Criteria:

* Contraindication to ESWL
* No interest in music listening
* < 18 years and > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
percentage of patients who appreciated music listening during SWL without anesthesia | 10 mins after SWL treatment completed
  patients were asked if they appreciated music listening during swl

SECONDARY OUTCOMES:
percentage of patients who considered music useful to relieve pain | 10 mins after SWL treatment completed
  patients were asked if they considered music useful to relieve pain during swl
change in SW voltage (kV) | 10 mins after SWL treatment completed
  change in SW voltage (kV)
change in VAS score | 10 mins after SWL treatment completed
  Visual analogue scale (VAS) - 0 to 10, higher values, worse pain
change in analgesic request | 10 mins after SWL treatment completed
  change in analgesic request
change in requested interruptions | 10 mins after SWL treatment completed
  change in requested interruptions
change on VAS scores separately measured in each part of the treatment | 10 mins after SWL treatment completed
  Visual analogue scale (VAS) - 0 to 10, higher values, worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Andrea MD Bosio, MD, Study Chair — AOU città dellaSalute e della Scienza, Torino; Andrea MD Bosio, MD, Principal Investigator — AOU città dellaSalute e della Scienza, Torino; Andrea MD Bosio, MD, Study Director — AOU città dellaSalute e della Scienza, Torino
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Italy